CLINICAL TRIAL: NCT00461760
Title: A Randomized Controlled Evaluation of HPV Testing for Cervical Cancer Screening
Brief Title: HPV Testing for Cervical Cancer Screening Study
Acronym: HPVFOCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Gina Ogilvie, Dr. Gina Ogilvie, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H06-04032
Record Dates: First submitted 2007-04-13; First posted 2007-04-18 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Cervical Cancer Screening
Keywords: HPV Screening/Testing for cervical cancer screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Women with normal cytology at recruitment will be recalled for their next routine screen at 2 years and if negative again, for their exit screen at 4 years, all according to current provincial guidelines.
  Interventions: Procedure: Cervical cancer screening undertaken by HPV testing as a single primary screening test with cytology triage of women who are HPV positive
- 2 (Active Comparator): Women with abnormal cytology at recruitment or at the 2 year screen will be followed according to provincial guidelines based on their cytology results.
  Interventions: Procedure: Cervical cancer screening undertaken by HPV testing as a single primary screening test with cytology triage of women who are HPV positive

INTERVENTIONS:
Procedure: Cervical cancer screening undertaken by HPV testing as a single primary screening test with cytology triage of women who are HPV positive — See Detailed Description.
  Arms: 1
Procedure: Cervical cancer screening undertaken by HPV testing as a single primary screening test with cytology triage of women who are HPV positive — See detailed description.
  Arms: 2

SUMMARY:
This is a randomised controlled trial of HPV testing with cytology triage for HPV positive women compared to liquid-based cervical cytology (LBC). Although LBC is not widely used for cervical cancer screening in Canada at present, the Pan-Canadian Cervical Cancer Forum has recommended its use and as it is likely to be the standard of care by the time these data are published, the trial has been designed to account for this. Further, LBC will improve the cost-effectiveness of HPV testing because the LBC medium is suitable for both HPV testing as well as cytology and thereby allows the triage testing to be undertaken from the same sample without having to recall the women.

DETAILED DESCRIPTION:
There is now an overwhelming body of data to show that HPV testing has the potential to improve the effectiveness of cervical cancer screening programs and thereby reduce rates of cervical cancer. As a result, there is a growing ethical dilemma in that we potentially have the means to prevent disease and death among Canadian women, and yet the studies that have been undertaken do not offer the standard of evidence that is required to change large-scale public health programs such as cervical cancer screening. In recognition of this, the Pan-Canadian Cervical Cancer Forum (PCCCF) has called for the evaluation of HPV testing within the context of a Canadian organised cervical cancer screening program. Given the potential health benefits that could be achieved, and that a pan-Canadian expert group has issued a consensus statement calling for the evaluation of HPV testing for primary screening, it is now an imperative that a properly designed and powered study be conducted to definitively establish whether it will provide the hypothesised health benefits within Canada.

The results of this trial will demonstrate whether or not the use of HPV testing as a single primary screening test within an organised Canadian cervical cancer screening program will be able to 1) provide further reductions in cervical cancer incidence, 2) allow the screening interval to be extended and 3) improve the cost-effectiveness of cervical cancer screening. If this trial demonstrates that HPV testing will provide these benefits, the BCCA will implement HPV testing as a single primary screening test within the provincial cervical cancer screening program and the trial will directly influence the provision of this service in BC. In addition, many other Canadian provinces and territories are either implementing or have plans to implement screening programs similar to the one in BC and by the time this trial is completed, many will have these programs operating. Therefore, the results of this trial will be directly applicable to these programs and constitute a demonstration project for the rest of Canada.

A list of women who are due for cervical screening will be sent to study collaborating Family Physicians (FPs) each month from the study centre in the provincial screening program. An invitation letter will be sent by the FP to potentially eligible women due for cervical cancer screening. If women are interested in participating, they will contact the study centre for more information. Study staff discuss the details of the trial with them, confirm eligibility and administer a short survey. Women who consent to the trial will visit the FP for their screening test and samples will be obtained and sent to the BC Central Laboratory Service (BC-CLS) where it will be randomized into one of the study arms:

Note: Recruitment to the safety arm was complete December 31, 2010 and from that point forward, women randomized 1:1 into the control or intervention arms only. A total of ~25,000 women (~9140 each in the Control and Intervention arms respectively, and ~6,000 in the Safety arm) will be enrolled in the FOCAL trial.

Control arm:

Sample tested with LBC.

* Those with negative results will be recalled for next screen at 2 years and if negative again, for the exit screen at 4 years. Those with positive cytology results have reflex HPV testing, or referral to colposcopy based on results.
* Exit screen testing is both HPV and cytology testing

  2-year safety-check arm: Sample tested for HPV.
* HPV negatives recalled at 2-years for the exit screen with cytology
* Women who are HPV positive will have their residual LBC specimen processed for cytology and be managed according to the same protocol as HPV-positive women in the 4-year intervention arm.

  4-year intervention arm: Sample tested for HPV.
* HPV negatives will be recalled at 4 years for their exit screen with HPV and cytology testing
* Women who are HPV positive will undergo reflex cytology testing and those cytology negative will be recalled at 12 months for HPV testing and cytology. At 12 mos, participants will be referred to colposcopy if > or =ASC-US or HPV positive. If HPV and cytology negative at 12 months returned to the routine screening pool for this arm and recalled for the exit screen at 4-years.
* Women who are HPV positive and > or = ASC-US will be referred to colposcopy and managed according to colposcopy results.

ELIGIBILITY:
Inclusion Criteria:

Women from 25 to 65 years of age, registered with the Medical Services Plain in BC attending a collaborating healthcare provider for routine cervical screening in Metro Vancouver or Greater Victoria.

Exclusion Criteria:

1. pregnant
2. history of invasive cervical cancer
3. no cervix
4. HIV positive or on immunosuppressive treatments
5. unable or unwilling to give informed consent
6. Treatment of moderate or greater dysplasia within last 5 years

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25223 (Actual)
Dates: Start 2007-03; Primary Completion 2017-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Histologically confirmed greater than or equal to CIN2 detected at 2 years in both the control and the safety-check arms. | 2 years
Histologically confirmed greater than or equal to CIN3 detected over the 4 years post recruitment in the control and intervention arms will be evaluated and compared as a surrogate marker for estimating reductions in the incidence of cervical cancer. | 4 years
Detection of histologically confirmed greater than or equal to CIN3 in the participants allocated to 6-month retesting.
The total estimated cost per woman screened and the total estimated cost per quality-adjusted life-year gained for each technology.

SECONDARY OUTCOMES:
Clearance of HPV infection in women who are HPV positive at recruitment
HPV type specific prevalence in the screening population

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Coldman, PhD, Principal Investigator — University of British Columbia; Gina Ogilvie, MD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Laurie Smith, Vancouver, British Columbia
  - BC Cancer, Vancouver, British Columbia
  - BC Center for Disease Control, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

REFERENCES:
- [Derived] Smith LW, Racey CS, Gondara L, Krajden M, Lee M, Martin RE, Stuart G, Peacock S, Coldman AJ, Franco EL, van Niekerk D, Ogilvie GS. Women's acceptability of and experience with primary human papillomavirus testing for cervix screening: HPV FOCAL trial cross-sectional online survey results. BMJ Open. 2021 Oct 7;11(10):e052084. doi: 10.1136/bmjopen-2021-052084. PMID 34620663